CLINICAL TRIAL: NCT07108153
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled Proof-of-concept Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of SION-719 When Added to Physician-prescribed Trikafta® in People With Cystic Fibrosis Who Are Homozygous for the F508del Mutation
Brief Title: Proof-of-concept Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of SION-719 When Added to Trikafta
Acronym: PreciSION CF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sionna Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SION-719-201
Record Dates: First submitted 2025-07-18; First posted 2025-08-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crossover Treatment Sequence 1: SION-719 followed by placebo-to-match SION-719 (Experimental): Participants receive SION-719 for one treatment period, and placebo to match SION-719 for the other treatment period. All participants will remain on their physician-prescribed Trikafta as background therapy throughout the study.
  Interventions: Drug: SION-719; Drug: Placebo-to-match SION-719
- Crossover Treatment Sequence 2: Placebo-to-match SION-719 followed by SION-719 (Experimental): Participants receive placebo to match SION-719 for one treatment period and SION-719 for the other treatment period. All participants will remain on their physician-prescribed Trikafta as background therapy throughout the study.
  Interventions: Drug: SION-719; Drug: Placebo-to-match SION-719

INTERVENTIONS:
Drug: SION-719 — All participants receive SION-719, as specified by their treatment sequence assignment
Drug: Placebo-to-match SION-719 — All participants receive placebo to match SION-719, as specified by their treatment sequence assignment

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of SION-719 when given to people with CF who are already taking Trikafta.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF with F508del homozygous genotype based on documented CFTR genotype laboratory report.
* Adherent to physician-prescribed Trikafta, as assessed by the Investigator, for at least 3 months prior to the Screening visit, taken at the recommended dose without modifications and on the regimen described in the current prescribing information.
* Stable CF disease without pulmonary exacerbation within 28 days before Baseline or acute non-CF-related illness within 14 days before Baseline.

Exclusion Criteria:

* Participant has clinically significant current or recurrent illness, other than CF
* Participant has a history of malignancy, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of recurrence for at least 1 year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of treatment emergent adverse events [Safety and Tolerability] when SION-719 is administered to people with cystic fibrosis (CF) who are taking a standard stable dose of physician-prescribed Trikafta | Day 1 through day 57
  Adverse events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE), v. 5.0

SECONDARY OUTCOMES:
Change from baseline in sweat chloride levels | Baseline to Day 15 in each treatment period
  Changes from baseline in sweat chloride levels will be analyzed with mixed model repeated measures (MMRM) methods.
Concentration of SION-719 in plasma and change of concentration of SION-719 in plasma. | Day 1 through day 57
  Concentrations of plasma SION-719 will be evaluated at each collected timepoint and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sionna Therapeutics Inc.
Locations (13):
- United States (10):
  - National Jewish Health, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - New York Medical College, Hawthorne, New York
  - Columbia University, New York, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Monash University, Melbourne, Victoria